CLINICAL TRIAL: NCT00577824
Title: Efficacy and Safety of LY2148568 in Japanese Patients With Type 2 Diabetes Who Are Treated With Oral Antidiabetic(s) But Not Well Controlled
Brief Title: Efficacy and Safety of Exenatide in Japanese Patients With Type 2 Diabetes Who Are Treated With Oral Antidiabetic(s)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H8O-JE-GWBB
Record Dates: First submitted 2007-12-18; First posted 2007-12-20 (Estimated); Results first posted 2009-12-31 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes
Keywords: diabetes; exenatide; LY2148568; Byetta; Lilly; Amylin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: exenatide
- 2 (Experimental)
  Interventions: Drug: exenatide
- 3 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: exenatide — subcutaneous injection, 5mcg, twice a day
  Other Names: LY2148568; Byetta
  Arms: 1
Drug: exenatide — subcutaneous injection, 10mcg, twice a day
  Other Names: LY2148568; Byetta
  Arms: 2
Drug: placebo — subcutaneous injection, volume equivalent to 5mcg or 10mcg exenatide, twice a day
  Arms: 3

SUMMARY:
This long term, placebo-controlled trial is intended to assess the efficacy and safety of exenatide, dosed twice a day, in Japanese patients with Type 2 Diabetes who are treated with oral antidiabetic(s) but not well controlled.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes.
* Has been treated by sulfonylurea (SU) alone, SU and biguanide, or SU and thiazolidinedione for at least 90 days prior to study start. In a patient receiving SU alone, the dose must be within the dose range from maximum maintenance dose to maximum approved dose. The patients with concomitant use of alpha glucosidase inhibitors (acarbose, voglibose or miglitol) or meglitinide derivatives (mitiglinide or nateglinide) can be included in this study, but these drugs must be discontinued at study start.
* Have HbA1c 7.0% to 10% at study start.
* Have a body weight >=50 kg.

Exclusion Criteria:

* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.
* Have participated in this study previously or any other study using exenatide or glucagon-like peptide-1 (GLP-1) analogs within the last 90 days.
* Have been treated with any exogenous insulin within 90 days before study start.
* Have been continuously treated with any drug that directly affects gastrointestinal motility for more than a total of 21 days in the 90 days prior to study start.
* The combination therapy of sulfonylurea, biguanide and thiazolidinedione is not allowed.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2008-01; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, MD, Study Director — Eli Lilly and Company
Locations (12):
- Japan (12):
  - Research Site, Chiba
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Hyōgo
  - Research Site, Ibaraki
  - Research Site, Kanagawa
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Nagano
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Tokyo

REFERENCES:
- [Result] Kadowaki T, Namba M, Imaoka T, Yamamura A, Goto W, Boardman MK, Sowa H. Improved glycemic control and reduced bodyweight with exenatide: A double-blind, randomized, phase 3 study in Japanese patients with suboptimally controlled type 2 diabetes over 24 weeks. J Diabetes Investig. 2011 Jun 5;2(3):210-7. doi: 10.1111/j.2040-1124.2010.00084.x. PMID 24843486
- [Result] Inagaki N, Ueki K, Yamamura A, Saito H, Imaoka T. Long-term safety and efficacy of exenatide twice daily in Japanese patients with suboptimally controlled type 2 diabetes. J Diabetes Investig. 2011 Nov 30;2(6):448-56. doi: 10.1111/j.2040-1124.2011.00137.x. PMID 24843529
- [Derived] Pencek R, Blickensderfer A, Li Y, Brunell SC, Anderson PW. Exenatide twice daily: analysis of effectiveness and safety data stratified by age, sex, race, duration of diabetes, and body mass index. Postgrad Med. 2012 Jul;124(4):21-32. doi: 10.3810/pgm.2012.07.2567. PMID 22913891
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- 5mcg Exenatide BID: exenatide SC 5mcg, twice daily
- 10mcg Exenatide BID: exenatide SC 10mcg, twice daily
- Placebo BID: placebo SC, twice daily
Period: Overall Study
Arm/Group | 5mcg Exenatide BID | 10mcg Exenatide BID | Placebo BID
Started | 72 (Started=Randomized) | 73 | 36
Full Analysis Set | 72 (Full Analysis Set=subject received at least one dose of study medication (active or placebo)) | 72 | 35
Completed | 65 | 53 | 34
Not Completed | 7 | 20 | 2
Not completed — Adverse Event | 6 | 18 | 1
Not completed — Patient decision | 0 | 1 | 1
Not completed — Protocol Violation | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 5mcg Exenatide BID | 10mcg Exenatide BID | Placebo BID | Total
Number analyzed (Participants) | 72 | 72 | 35 | 179
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 53 | 46 | 27 | 126
  >=65 years | 19 | 26 | 8 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (9.33) | 59.4 (9.75) | 56.3 (11.41) | 58.4 (9.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 11 | 57
  Male | 49 | 49 | 24 | 122

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Hemoglobin (HbA1c) From Baseline to Week 24
Description: Change in HbA1c from baseline following 24 weeks of treatment (i.e., HbA1c at week 24 minus HbA1c at week 0)
Time Frame: baseline, 24 weeks
Population: Full analysis set; Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: Percentage of hemoglobin
Arm/Group | 5mcg Exenatide BID | 10mcg Exenatide BID | Placebo BID
Number analyzed (Participants) | 71 | 72 | 35
Percentage of hemoglobin | -1.34 (0.11) | -1.62 (0.11) | -0.28 (0.15)
Statistical Analysis 1: Comparison: 10mcg Exenatide BID vs Placebo BID; Test type: Superiority or Other; p < 0.001, ANCOVA — Bonferroni's method was used to adjustment for multiplicity, and significant level was set to 2.5%(two-sided); ANCOVA model with treatment group as a factor and baseline value as the covariate

2. Secondary Outcome: Percentage of Patients Achieving HbA1c < 7.0%
Description: Percentage of subjects whose HbA1c was >=7.0% at baseline who achieved an HbA1c < 7.0% at endpoint (i.e., number of eligible subjects who achieved HbA1c < 7.0% divided by total number of eligible subjects times 100)
Time Frame: 24 weeks
Population: Full analysis set; Last observation carried forward. Only those patients with HbA1c >=7% at baseline included.
Measure: Number; unit: percentage of participants
Arm/Group | 5mcg Exenatide BID | 10mcg Exenatide BID | Placebo BID
Number analyzed (Participants) | 70 | 69 | 33
percentage of participants | 67.1 | 71.0 | 15.2
Statistical Analysis 1: Comparison: 5mcg Exenatide BID vs 10mcg Exenatide BID vs Placebo BID; Test type: Superiority or Other; p < 0.001, Cochran-Armitage

3. Secondary Outcome: Percentage of Patients Achieving HbA1c < 6.5%
Description: Percentage of subjects whose HbA1c was >=6.5% at baseline who achieved an HbA1c < 6.5% at endpoint (i.e., number of eligible subjects who achieved HbA1c < 6.5% divided by total number of eligible subjects times 100)
Time Frame: 24 weeks
Population: Full analysis set; Last observation carried forward. Only subjects whose HbA1c was >=6.5% at baseline were included.
Measure: Number; unit: percentage of participants
Arm/Group | 5mcg Exenatide BID | 10mcg Exenatide BID | Placebo BID
Number analyzed (Participants) | 71 | 72 | 35
percentage of participants | 36.6 | 47.2 | 8.6
Statistical Analysis 1: Comparison: 5mcg Exenatide BID vs 10mcg Exenatide BID vs Placebo BID; Test type: Superiority or Other; p < 0.001, Cochran-Armitage

4. Secondary Outcome: Change in Fasting Blood Glucose
Description: Change in fasting blood glucose from baseline to endpoint (i.e., fasting blood glucose at week 24 minus fasting blood glucose at week 0)
Time Frame: baseline, week 24
Population: Full analysis set; Last observation carried forward
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | 5mcg Exenatide BID | 10mcg Exenatide BID | Placebo BID
Number analyzed (Participants) | 71 | 72 | 35
mg/dL | -25.1 (3.83) | -29.0 (3.81) | -7.6 (5.46)
Statistical Analysis 1: Comparison: 10mcg Exenatide BID vs Placebo BID; Test type: Superiority or Other; p < 0.002, ANCOVA — No adjustment for multiplicity. Significance level was 5% (two-sided)

5. Secondary Outcome: Change in Body Weight
Description: Change in body weight form baseline to endpoint (i.e., body weight at week 24 minus body weight at week 0)
Time Frame: baseline, week 24
Population: Full analysis set; Last observation carried forward
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | 5mcg Exenatide BID | 10mcg Exenatide BID | Placebo BID
Number analyzed (Participants) | 71 | 72 | 35
kg | -0.39 (0.28) | -1.54 (0.27) | -0.47 (0.39)
Statistical Analysis 1: Comparison: 10mcg Exenatide BID vs Placebo BID; Test type: Superiority or Other; p = 0.026, ANCOVA — No adjustment for multiplicity. Significance level was 5% (two-sided)

6. Secondary Outcome: Change in Total Cholesterol
Description: Change in total cholesterol from baseline to endpoint (i.e., total cholesterol at week 24 minus total cholesterol at week 0)
Time Frame: baseline, week 24
Population: Full analysis set; Last observation carried forward
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | 5mcg Exenatide BID | 10mcg Exenatide BID | Placebo BID
Number analyzed (Participants) | 71 | 72 | 35
mg/dL | -14.45 (3.36) | -7.01 (3.13) | -4.80 (3.76)
Statistical Analysis 1: Comparison: 10mcg Exenatide BID vs Placebo BID; Test type: Superiority or Other; p = 0.672, t-test, 2 sided

7. Secondary Outcome: Change in Low Density Lipoprotein Cholesterol (LDL-C)
Description: Change in LDL-C from baseline to endpoint (i.e., LDL-C at week 24 minus LDL-C at week 0)
Time Frame: baseline, week 24
Population: Full analysis set; Last observation carried forward.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | 5mcg Exenatide BID | 10mcg Exenatide BID | Placebo BID
Number analyzed (Participants) | 71 | 72 | 35
mg/dL | -8.89 (3.01) | -5.03 (2.45) | -2.66 (3.50)
Statistical Analysis 1: Comparison: 10mcg Exenatide BID vs Placebo BID; Test type: Superiority or Other; p = 0.580, t-test, 2 sided

8. Secondary Outcome: Change in High Density Lipoprotein Cholesterol (HDL-C)
Description: Change in HDL-C from baseline to endpoint (i.e., HDL-C at week 24 minus HDL-C at week 0)
Time Frame: baseline, week 24
Population: Full analysis set; Last observation carried forward.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | 5mcg Exenatide BID | 10mcg Exenatide BID | Placebo BID
Number analyzed (Participants) | 71 | 72 | 35
mg/dL | -4.63 (0.91) | -4.22 (0.70) | -0.97 (1.20)
Statistical Analysis 1: Comparison: 10mcg Exenatide BID vs Placebo BID; Test type: Superiority or Other; p = 0.014, t-test, 2 sided

9. Secondary Outcome: Change in Triglycerides
Description: Change in triglycerides from baseline to endpoint (i.e., triglycerides at week 24 minus triglycerides at week 0)
Time Frame: baseline, week 24
Population: Full analysis set; Last observation carried forward
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | 5mcg Exenatide BID | 10mcg Exenatide BID | Placebo BID
Number analyzed (Participants) | 71 | 72 | 35
mg/dL | 4.00 (15.59) | 4.13 (8.03) | -4.60 (7.25)
Statistical Analysis 1: Comparison: 10mcg Exenatide BID vs Placebo BID; Test type: Superiority or Other; p = 0.490, t-test, 2 sided

10. Secondary Outcome: Change in Waist Size
Description: Change in waist size from baseline to endpoint (i.e., waist size at week 24 minus waist size at week 0)
Time Frame: baseline, week 24
Population: Full Analysis Set; Last Observation Carried Forward
Measure: Mean (Standard Error); unit: cm
Arm/Group | 5mcg Exenatide BID | 10mcg Exenatide BID | Placebo BID
Number analyzed (Participants) | 70 | 71 | 35
cm | -0.17 (0.36) | -1.81 (0.46) | 0.41 (0.45)
Statistical Analysis 1: Comparison: 10mcg Exenatide BID vs Placebo BID; Test type: Superiority or Other; p = 0.003, t-test, 2 sided

11. Secondary Outcome: Change in Waist-to-hip Ratio
Description: Change in waist-to-hip ratio from baseline to endpoint (i.e., waist-to-hip ratio at week 24 minus waist-to-hip ratio at week 0). Waist-to-hip ratio is waist circumference divided by hip circumference.
Time Frame: baseline, week 24
Population: Full Analysis Set; Last Observation Carried Forward
Measure: Mean (Standard Error); unit: ratio (cm/cm)
Arm/Group | 5mcg Exenatide BID | 10mcg Exenatide BID | Placebo BID
Number analyzed (Participants) | 70 | 71 | 35
ratio (cm/cm) | 0.0016 (0.0047) | -0.0108 (0.0047) | -0.0007 (0.0061)
Statistical Analysis 1: Comparison: 10mcg Exenatide BID vs Placebo BID; Test type: Superiority or Other; p = 0.208, t-test, 2 sided

12. Secondary Outcome: 7 Point Self-monitored Blood Glucose (SMBG) Profiles at Baseline and Week 24
Description: Self-monitored blood glucose at 7 different time points during the day (glucose measurements before and 2 hours after the start of the morning, midday, and evening meals, and at bedtime).
Time Frame: baseline, week 24
Population: Full Analysis Set; Last Observation Carried Forward
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 5mcg Exenatide BID | 10mcg Exenatide BID | Placebo BID
Number analyzed (Participants) | 72 | 71 | 35
mg/dL
  30 minutes prior to breakfast SMBG at week 0 | 169 (36.3) | 175 (40.9) | 170 (38.6)
  30 minutes prior to breakfast SMBG at week 24 | 150 (36.4) | 140 (32.2) | 167 (37.9)
  2hr post-breakfast SMBG at week 0 | 261 (50.5) | 263 (55.1) | 254 (65.1)
  2hr post-breakfast SMBG at week 24 | 178 (61.1) | 149 (54.4) | 257 (74.5)
  30 minutes prior to lunch SMBG at week 0 | 179 (48.4) | 189 (68.4) | 179 (49.2)
  30 minutes prior to lunch SMBG at week 24 | 155 (43.9) | 152 (41.3) | 182 (57.0)
  2hr post-lunch SMBG at week 0 | 263 (62.7) | 268 (62.4) | 264 (51.7)
  2hr post-lunch SMBG at week 24 | 213 (63.2) | 195 (60.7) | 254 (73.5)
  30 minutes prior to dinner SMBG at week 0 | 166 (53.7) | 176 (51.4) | 173 (42.5)
  30 minutes prior to dinner SMBG at week 24 | 149 (45.1) | 140 (35.5) | 181 (57.0)
  2hr post-dinner SMBG at week 0 | 246 (53.4) | 247 (63.6) | 239 (49.1)
  2hr post-dinner SMBG at week 24 | 160 (62.8) | 141 (57.7) | 247 (78.6)
  bedtime SMBG at week 0 | 216 (53.7) | 225 (66.2) | 206 (46.8)
  bedtime SMBG at week 24 | 170 (48.9) | 151 (44.3) | 212 (63.5)

13. Secondary Outcome: Change in Homeostasis Model Assessment - Beta Cell Function (HOMA-B)
Description: Change in HOMA-B from baseline to endpoint (i.e., HOMA-B at week 24 minus HOMA-B at week 0). HOMA-B is a measurement of beta cell function.
Time Frame: baseline, week 24
Population: Full Analysis Set; Last Observation Carried Forward
Measure: Mean (Standard Error); unit: ratio
Arm/Group | 5mcg Exenatide BID | 10mcg Exenatide BID | Placebo BID
Number analyzed (Participants) | 70 | 72 | 35
ratio | 2.475 (10.566) | 6.836 (13.858) | -0.707 (3.436)
Statistical Analysis 1: Comparison: 10mcg Exenatide BID vs Placebo BID; Test type: Superiority or Other; p = 0.708, t-test, 2 sided

14. Secondary Outcome: Change in Homeostasis Model Assessment - Insulin Resistance (HOMA-R)
Description: Change in HOMA-R from baseline to endpoint (i.e., HOMA-R at week 24 minus HOMA-R at week 0). HOMA-R is a measurement of insulin resistance.
Time Frame: baseline, week 24
Population: Full Analysis Set; Last Observation Carried Forward
Measure: Mean (Standard Error); unit: ratio
Arm/Group | 5mcg Exenatide BID | 10mcg Exenatide BID | Placebo BID
Number analyzed (Participants) | 70 | 72 | 35
ratio | -0.541 (0.402) | -0.366 (0.188) | -0.375 (0.164)
Statistical Analysis 1: Comparison: 10mcg Exenatide BID vs Placebo BID; Test type: Superiority or Other; p = 0.974, t-test, 2 sided

15. Secondary Outcome: Change in Serum Insulin
Description: Change in serum insulin from baseline to endpoint (i.e., serum insulin at week 24 minus serum insulin at week 0)
Time Frame: baseline, week 24
Population: Full Analysis Set; Last Observation Carried Forward
Measure: Mean (Standard Deviation); unit: mcU/mL
Arm/Group | 5mcg Exenatide BID | 10mcg Exenatide BID | Placebo BID
Number analyzed (Participants) | 72 | 72 | 35
mcU/mL | -0.2 (5.03) | 0.2 (3.42) | -0.7 (2.42)

16. Secondary Outcome: Change in C-peptide
Description: Change in C-peptide from baseline to endpoint (i.e., C-peptide at week 24 minus C-peptide at week 0)
Time Frame: baseline, week 24
Population: Full Analysis Set; Last Observation Carried Forward
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | 5mcg Exenatide BID | 10mcg Exenatide BID | Placebo BID
Number analyzed (Participants) | 70 | 72 | 35
ng/mL | 0.05 (0.11) | 0.07 (0.07) | -0.08 (0.06)
Statistical Analysis 1: Comparison: 10mcg Exenatide BID vs Placebo BID; Test type: Superiority or Other; p = 0.200, t-test, 2 sided

17. Secondary Outcome: Change in 1,5-anhydroglucitol
Description: Change in 1,5-anhydroglucitol from baseline to endpoint (i.e., 1,5-anhydroglucitol at week 24 minus 1,5-anhydroglucitol at week 0)
Time Frame: baseline, week 24
Population: Full Analysis Set; Last Observation Carried Forward
Measure: Mean (Standard Error); unit: mcg/mL
Arm/Group | 5mcg Exenatide BID | 10mcg Exenatide BID | Placebo BID
Number analyzed (Participants) | 64 | 66 | 32
mcg/mL | 5.29 (0.55) | 4.52 (0.54) | 0.66 (0.30)
Statistical Analysis 1: Comparison: 10mcg Exenatide BID vs Placebo BID; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Up to 30 weeks (Up to a 6 week screening period, and then 24 weeks on treatment).
Arm/Group | 5mcg Exenatide BID | 10mcg Exenatide BID | Placebo BID
Serious Adverse Events (participants affected / at risk) | 2/72 | 0/72 | 4/35
Other Adverse Events (participants affected / at risk) | 63/72 | 63/72 | 22/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 5mcg Exenatide BID (N=72) | 10mcg Exenatide BID (N=72) | Placebo BID (N=35)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Gastric mucosal lesion (Gastrointestinal disorders) | 0 | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Major depression (Psychiatric disorders) | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Sleep apnea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 5mcg Exenatide BID (N=72) | 10mcg Exenatide BID (N=72) | Placebo BID (N=35)
Hypoglycemia (Metabolism and nutrition disorders) | 37 | 42 | 8
Nausea (Gastrointestinal disorders) | 18 | 26 | 3
Blood glucose decreased (Investigations) | 10 | 18 | 4
Vomiting (Gastrointestinal disorders) | 3 | 12 | 1
Constipation (Gastrointestinal disorders) | 10 | 11 | 1
Nasopharyngitis (Infections and infestations) | 8 | 9 | 8
Stomach discomfort (Gastrointestinal disorders) | 7 | 9 | 1
Decreased appetite (Metabolism and nutrition disorders) | 7 | 9 | 1
Anorexia (Metabolism and nutrition disorders) | 2 | 8 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 5 | 0
Diarrhoea (Gastrointestinal disorders) | 8 | 4 | 2
Feeling abnormal (General disorders) | 0 | 4 | 0
Malaise (General disorders) | 2 | 4 | 2
Blood creatinine phosphokinase increased (Investigations) | 0 | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 3 | 2 | 2
Bronchitis (Infections and infestations) | 1 | 2 | 2
Eczema (Skin and subcutaneous tissue disorders) | 4 | 2 | 0
Headache (Nervous system disorders) | 4 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days